CLINICAL TRIAL: NCT06306313
Title: Effects of Robot-Assisted Rehabilitation on Upper Extremity Functions and Activities of Daily Living in Chronic Stroke Patients
Brief Title: Effects of Robot-Assisted Rehabilitation on Upper Extremity Functions in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fatih Tekin, Assist. Prof., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ReoGo
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Upper Extremity Paresis
Keywords: Robotic Rehabilitation; Chronic Stroke; Upper Limb; Activities of Daily Living
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Conventional physiotherapy will be applied in a single session of 45 minutes a day, 3 days a week for 4 weeks, and in addition, robot-assisted therapy will be applied with the ReoGo Upper Extremity Exoskeleton Robot in a single session of 60 minutes a day, 5 days a week for 4 weeks. Evaluations will be made at the beginning and end of the treatment process.
  Interventions: Device: ReoGo; Other: Conventional Physiotherapy
- Control Group (Active Comparator): The control group will receive only conventional physiotherapy in a single session of 45 minutes a day, 3 days a week for 4 weeks. Evaluations will be made at the beginning and end of the treatment process.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Device: ReoGo — ReoGo is a fixed arm rehabilitation exoskeleton that comes on a small and compact wheeled platform. The end-effector extension is capable of producing a wide range or repeatable movements in 3D space. ReoGo can be used by both adults and children. It is an arm rehabilitation exoskeleton with a fixed base. Its design allows limited controlled movements of the shoulder as well as the elbow and wrist.
  Arms: Experimental
Other: Conventional Physiotherapy — Physiotherapy protocols will be created with traditional physiotherapy practices such as neurodevelopmental techniques based on muscle strengthening and task-oriented exercises. Protocols in general terms; It will include passive and active joint range of motion exercises, stretching exercises, stimulation and facilitation techniques, strengthening exercises, fine motor skills and functional task training for daily living activities. Protocols will be tailored to each patient's level of motor impairment and functional needs.

SUMMARY:
The most common problem caused by stroke is motor activity limitation that reduces muscle movement and mobility. But stroke can also lead to sensory and cognitive impairment. Additionally, the ability to independently carry out activities of daily living and participate in social and community life is greatly reduced. Up to 85% of stroke patients experience hemiparesis immediately after stroke, while 55% to 75% of survivors continue to experience reduced quality of life with motor impairments.

It requires long-term physical rehabilitation to achieve functional recovery in the upper extremity, maximum independence and the highest possible quality of life. Different methods can be used to achieve these results, but there is no clear evidence yet as to which treatment method gives the best results. Scientific evidence shows that a multifactorial approach and high-intensity treatment accelerates the motor recovery of the upper extremities in stroke rehabilitation. Passive and active upper extremity movements appear to increase motor recovery due to their effects on somatosensory input, motor planning, soft tissue properties and spasticity.

In recent years, robotic devices have emerged that have been proven to improve the motor performance of the upper extremity in chronic stroke patients. There are also studies showing that robotic device-assisted upper extremity therapy can contribute to the development of sensorimotor skills in plegic patients. However, in the current literature, there is still a need for randomized controlled studies in this field. The aim of this study is to investigate the effects of robot-assisted therapy on upper extremity functions and daily living activities in the rehabilitation of chronic stroke patients. After the demographic data of the cases in both groups are obtained, evaluations will be made before the study. Then, the study group will receive conventional physiotherapy in a single session of 45 minutes a day, 3 days a week for 4 weeks, and in addition robot-assisted therapy with the ReoGo Upper Extremity Exoskeleton Robot in a single session of 60 minutes a day, 5 days a week for 4 weeks. The control group will receive only conventional physiotherapy in a single session of 45 minutes a day, 3 days a week for 4 weeks. The initial evaluations will be repeated after the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Having had a single stroke
* Having had at least 6 months since the stroke
* Having hemiparesis/hemiplegia following the stroke
* Having mental health sufficient to meet all evaluation and treatment procedures in the study

Exclusion Criteria:

* Having a history of disease other than stroke that affects the use of the upper extremity

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Upper Extremity Evaluation Scale | Through study completion, an average of 3 months
  It is a scale based on measuring performance and is frequently recommended for use especially in stroke patients. Test; It consists of subsections: reflex activity, flexor and extensor synergy, combined synergistic movements, non-synergistic movements, normal reflex activity, wrist and hand evaluation, coordination and speed evaluation. It consists of 33 items in total and each item is scored between 0 and 2 points (0: cannot do, 1: partially can, 2: completely can). Total score is 66. It is easy to apply, does not require a lot of equipment, items found at home are sufficient and takes about 30 minutes.
Functional Independence Scale | Through study completion, an average of 3 months
  It is used to evaluate the independence of patients in daily living activities. It has 13 items consisting of 4 subcategories to evaluate motor functional limitation, including self-care, sphincter control, transfer and displacement. To evaluate cognitive functional limitation, it has 5 items consisting of 2 subcategories including communication and social perception. It is a scale divided into 6 categories and consisting of 18 items in total. Each item is rated on a 7-point scale. A score of 7 indicates complete independence, while a score of 1 indicates maximum dependence. The lowest score that can be obtained from the scale is 18 and the highest score is 126. As the score obtained from the scale increases, the patient's level of independence increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No